CLINICAL TRIAL: NCT06845410
Title: Clinical Features, Current Treatment and Clinical Outcomes in Patients With Inflammation-associated Non-rapidly-progressive Coronary Artery Disease (INR-CAD): a Cohort Study
Brief Title: Clinical Features, Current Treatment and Clinical Outcomes in Patients With INR-CAD: a Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Other Study IDs: K6722
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease Progression; Coronary Artery Stenosis; Coronary Artery Restenosis; Inflammation; Inflammatory Disease; Inflammation Vascular
Keywords: Coronary Artery Disease; Progression, Disease; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis; Inflammation; Disease Progression | interventions — Secondary Prevention; Immunosuppression Therapy; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood samples will be retained for potential RNA sequencing, proteomics, and metabolomics studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INR-CAD Group: Patients who have been clinically diagnosed as INR-CAD and received, or are receiving, or will receive the 24-month clinical follow-up according to the clinical diagnostic criteria and follow-up protocol for INR-CAD.
  Interventions: Behavioral: Healthy life style; Drug: Secondary prevention for atherosclerotic coronary artery disease; Drug: Immunosuppressive Therapy; Procedure: Coronary revascularization; Drug: Supportive therapies

INTERVENTIONS:
Behavioral: Healthy life style — Healthy diet, regular exercise, and quitting smoking
Drug: Secondary prevention for atherosclerotic coronary artery disease — Antiplatelet therapy, as well as medications for control of heart rate, blood pressure, low-density lipoprotein cholesterol, and blood glucose
Drug: Immunosuppressive Therapy — Glucocorticoids and/or immunosuppressive agents
Procedure: Coronary revascularization — Percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG).
Drug: Supportive therapies — Medical interventions for prevention and treatment of the side effects of the above treatment, such as abnormal liver function, hypocalcemia, hypokalemia, peptic ulcer, infection, et al.

SUMMARY:
This is a cohort study to investigate the clinical features, current treatment and clinical outcomes in patients with inflammation-associated non-rapidly-progressive coronary artery disease (INR-CAD).

DETAILED DESCRIPTION:
A special type of coronary artery disease (CAD) has been identified in our clinical practice. The patients have significantly different clinical features from those of typical atherosclerotic coronary artery disease (AS-CAD), including: 1) predominantly female; 2) early onset CAD; 3) lack of traditional atherosclerotic risk factors; 4) often with evidence of chronic inflammation; 5) responding poorly to intensified secondary prevention and optimized coronary revascularization (percutaneous coronary intervention [PCI] or coronary bypass graft [CABG]); 6) delayed disease progression on immunosuppressive therapy. This special type of CAD is named with inflammation-associated coronary artery disease (I-CAD). Currently, the pathogenesis as well as the optimal approach regarding the diagnosis and treatment of I-CAD remain unknown.

Based on the rate of disease progression and the urgency for clinical management, I-CAD is classified into two categories: 1) inflammation-associated rapidly-progressive coronary artery disease (IR-CAD), which is defined as I-CAD with progression of coronary de novo and/or restenotic lesions within 6 months or within 12 months (only for patients receiving immunosuppressive therapy within 24 months); 2) inflammation-associated non-rapidly-progressive coronary artery disease (INR-CAD), which is defined as I-CAD not fulfilling the criteria for IR-CAD.

It has been recognized in our clinical practice that INR-CAD is a highly heterogeneous group of diseases. Therefore, the present observational cohort study was designed to investigate the clinical features, current treatment and clinical outcomes in patients with INR-CAD.

All patients who have been admitted to the Department of Cardiology, Peking Union Medical College Hospital (PUMCH) since January 1, 2022 will be screened for study participation. Clinical diagnostic criteria and a clinical follow-up protocol have been specifically designed for INR-CAD in our center. Patients are clinically diagnosed as INR-CAD if they 1) have angiographic evidence of coronary lesions (de novo or restenotic); 2) have evidence of chronic inflammation (positive inflammatory markers or positive autoantibodies or established diagnosis of chronic inflammatory diseases or use of immunosuppressive therapy) within 24 months; 3) not meet the clinical diagnostic criteria for IR-CAD. Once the clinical diagnosis is established, INR-CAD patients will receive a 24-month clinical follow-up according to the clinical follow-up protocol for INR-CAD in PUMCH. Patients who have been clinically diagnosed as INR-CAD and received, or are receiving, or will receive the 24-month clinical follow-up will be enrolled in the present cohort study.

The primary efficacy endpoint is major adverse cardiovascular events (MACE). The secondary efficacy endpoints include the individual components of MACE, exercise capacity, angiographic metrics of coronary lesions, and inflammatory markers. The safety endpoints are major bleeding events and severe infection events.

For the endpoints which are categorical variables, e.g., MACE, the event rate for the first occurrence of each endpoint during the 24-month clinical follow-up will be calculated. Chi-square test or Fisher's exact test will be used to compare the event rate for each endpoint between patients with different diagnosis and/or those receiving different treatment, including patients 1) with vs. without established diagnosis of chronic inflammatory diseases; 2) receiving vs. not receiving immunosuppressive therapy; 3) receiving vs. not receiving coronary revascularization.

For the endpoints which are continuous variables, e.g., inflammatory markers, 1) paired t-test or paired rank sum test will be used to compare the level of each endpoint at the end of the 24-month clinical follow-up with that at baseline (the diagnosis of INR-CAD); 2) analysis of co-variance (ANCOVA) will be used to compare the level of each endpoint at the end of the 24-month clinical follow-up between patients with different diagnosis and/or those receiving different treatment, including patients ① with vs. without established diagnosis of chronic inflammatory diseases; ② receiving vs. not receiving immunosuppressive therapy; ③ receiving vs. not receiving coronary revascularization.

ELIGIBILITY:
Inclusion criteria

1. 18 years of age or older, male or female.
2. Negative results of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).
3. Meeting the clinical diagnostic criteria for INR-CAD, including: (1) Angiographic evidence of coronary lesions (≥ 50% diameter stenosis, de novo or restenotic); (2) Evidence of chronic inflammation within 24 months: (A) Positive inflammatory markers (erythrocyte sedimentation rate [ESR], high-sensitivity C-reactive protein [hs-CRP], interleukin-6 [IL-6], tumor necrosis factor-alpha [TNF-α], et al; at least twice, ≥ 12 weeks apart), or (B) Positive autoantibodies (at least twice, ≥ 12 weeks apart), or (C) Established diagnosis of chronic inflammatory diseases (autoimmune disease, systemic vasculitis, psoriasis, tuberculosis, et al), or (D) Receiving immunosuppressive therapy (glucocorticoids, immunosuppressive agents, et al).
4. NOT meeting the clinical diagnostic criteria for IR-CAD, including: (1) Hospitalization due to myocardial ischemia, including: (A) Typical symptoms of angina (Canadian Cardiovascular Society [CCS] III-IV), and (B) Non-invasive evidence of myocardial ischemia; (2) Angiographic evidence of new or worsened coronary lesions (de novo or restenotic) considered relevant to myocardial ischemia, which occurred: (A) Within 6 months of last coronary angiography in any patients, or (B) Within 12 months of last coronary angiography in patients receiving immunosuppressive therapy within 24 months.
5. Received, or are receiving, or will receive the 24-month clinical follow-up defined by the clinical follow-up protocol for INR-CAD.

Exclusion Criteria:

1. Other moderate to severe heart diseases (congenital heart disease, valvular heart disease, myocarditis, cardiomyopathy, pericardial diseases, pulmonary hypertension, heart failure, arrhythmia, et al).
2. Active malignancy (diagnosed within 12 months or with ongoing requirement for treatment).
3. Vital organ failure.
4. Life expectancy < 1 year.
5. In pregnancy or breast-feeding, or with intention to be pregnant during the study period.
6. Risk of non-compliance (history of drug addiction or alcohol abuse, et al).
7. Previous enrollment in this study.
8. Participation in another study within 30 days.
9. Involvement in the planning and conduct of this study (applying to investigators, contract research organization staffs, study site staffs, et al).
10. Any condition, which in the opinion of the investigators, would make it unsuitable for the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been admitted to the Department of Cardiology, Peking Union Medical College Hospital (PUMCH) since January 1, 2022 will be screened for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  The composite endpoint including death, or Q-wave myocardial infarction, or unplanned myocardial ischemia-driven coronary revascularization (PCI or CABG), or unplanned myocardial ischemia-driven hospitalization.

SECONDARY OUTCOMES:
Death | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  All-cause death.
Q-wave myocardial infarction | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  Myocardial injury due to myocardial ischemia, resulting in newly formed pathological Q waves in ≥ 2 contiguous leads or equivalent manifestations on electrocardiogram.
Unplanned myocardial ischemia-driven coronary revascularization | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  Unplanned coronary revascularization (PCI or CABG) due to myocardial ischemia.
Unplanned myocardial ischemia-driven hospitalization | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  Unplanned hospitalization due to myocardial ischemia.
Walking distance in 6 minutes | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of 6-minute walk test (6MWT).
Target lesion minimal lumen area (TL-MLA) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The minimum lumen area of the target lesion on optical coherence tomography (OCT).
Target lesion percent area stenosis (TL-%AS) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  Percent area stenosis (% AS) = { [ ( proximal RLA + distal RLA ) - (MLA × 2) ] / ( proximal RLA + distal RLA ) } × 100% in the cross-section with the MLA of the target lesion on optical coherence tomography (OCT). RLA = reference lumen area; MLA = minimum lumen area; % AS = percent area stenosis.
SYNTAX score | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of SYNTAX score calculation.
Number of vessel segments with coronary lesions | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  Number of vessel segments with diameter stenosis ≥ 50% on coronary angiogram.
Erythrocyte sedimentation rate (ESR) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of erythrocyte sedimentation rate (ESR) test.
High-sensitivity C-reactive protein (hs-CRP) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of serum high-sensitivity C-reactive protein (hs-CRP) test.
Interleukin-6 (IL-6) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of serum interleukin (IL)-6 test.
Tumor necrosis factor-alpha (TNF-α) | At the beginning (diagnosis of INR-CAD) and the end of the 24-month clinical follow-up.
  The result of serum tumor necrosis factor-alpha (TNF-α) test.

OTHER OUTCOMES:
Major bleeding events | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  Major bleeding events evaluated according to the Bleeding Academic Research Consortium (BARC) criteria.
Severe infection events | From the beginning (diagnosis of INR-CAD) to the end of the 24-month clinical follow-up.
  Infection events involving vital organs, or with complications (such as structural change and/or dysfunction of vital organs, septic shock, et al), or requiring hospitalization, or requiring treatment with intravenous antibiotics, or requiring treatment with interventional procedures or surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China